CLINICAL TRIAL: NCT05713981
Title: The Impact of Dry Eye Syndrome on Novel Metrics of Low Contrast Vision Before and After Therapeutic Meibomian Gland Expression
Brief Title: The Impact of Dry Eye Syndrome on Metrics of Low Contrast Vision Before and After Meibomian Gland Expression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Incarnate Word (Other)
Responsible Party: Principal Investigator, JEFFREY CARL RABIN, Professor and Assistant Dean for Graduate Studies, Research and Assessment and Chief, Visual Neurophysiology Service, University of the Incarnate Word
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-1283-EXP
Record Dates: First submitted 2022-12-29; First posted 2023-02-06 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Gene Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- non-invasive Meibomian gland (MG) expression (Experimental): Baseline testing of visual acuity, contrast sensitivity, color vision, and Innova, Inc. cone and B/W low contrast vision will be measured.
  The intervention will be standard clinical expression of Meibomian superior and inferior glands (MG) using a sterile cotton tip applicator to apply gentle pressure in a rolling motion in the direction of the MGs along the upper and lower eyelid margins to allow oil secretion of the tested eye. One drop of sterile saline will be instilled following the intervention to remove debris. The subject's visual acuity, contrast sensitivity, color vision, and Innova, Inc. cone and B/W low contrast vision will be measured before and after this intervention.
  Interventions: Procedure: Meibomian gland (MG) expression

INTERVENTIONS:
Procedure: Meibomian gland (MG) expression — The procedure is performed with a sterile cotton tip applicator once in the upper and lower eyelids of the subject's choosing.

SUMMARY:
The study aims to determine the impact of Meibomian Gland Dysfunction (MGD) dry eye on low contrast black/white (luminance) and cone color sensitivity performance and improvement in these functions after in-house non-invasive Meibomian gland (MG) expression.

DETAILED DESCRIPTION:
This study offers possible benefits from gland expression to patients and subjects in terms of clinical measurements and care associated with meibomian gland dysfunction impacting all age ranges. Prior studies show that these interventions improve dry eye symptoms with intent to improve vision, low contrast color, and B/W vision after intervention in this study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 18 years
* Healthy individuals with reported symptoms of dry eye such as burning, stinging, fluctuating vision, inappropriate tearing, and feelings of grittiness particularly with prolonged near work

Exclusion Criteria:

* Under the age of 18
* Individuals currently using prescription eye medications for dry eye / MGD / inflammation / Infections or any other treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Change in Cone Contrast Sensitivity on the Cone Contrast Test (CCT, Innova Systems, Inc.) | This test will occur prior to the intervention (Meibomian gland expression) and immediately after this intervention.
  This computer test measures the lowest contrast (contrast sensitivity) to see red, green and blue cone specific letters.
Change in Response Time on Cone Contrast Test (CCT, Innova Systems, Inc.) | This test will occur prior to the intervention (Meibomian gland expression) and immediately after this intervention.
  This computer test measures average response time in seconds to see red, green and blue low contrast letters.

SECONDARY OUTCOMES:
Change in Black White Contrast Sensitivity (Innova Systems, Inc) | This test will occur prior to the intervention (Meibomian gland expression) and immediately after this intervention.
  This computer test measures the lowest contrast (contrast sensitivity) to see black/white letters.
Change in Response Time on Black White Contrast Sensitivity Test (Innova Systems, Inc) Response Time | This test will occur prior to the intervention (Meibomian gland expression) and immediately after this intervention.
  This computer test measures average response time in seconds to see low contrast black/white letters
Change in Visual Acuity Test at Low Contrast (Innova Systems, Inc) | This test will occur prior to the intervention (Meibomian gland expression) and immediately after this intervention.
  This computer test measures the smallest low contrast letters which can be seen.
Change in Response Time on Visual Acuity Test at Low Contrast (Innova Systems, Inc) | This test will occur prior to the intervention (Meibomian gland expression) and immediately after this intervention.
  This computer test measures average response time in seconds to see low contrast visual acuity letters
Change in Sensitivity on Cone Contrast Color Naming test (CCNT) | This test will occur prior to the intervention (Meibomian gland expression) and immediately after this intervention.
  This computer test measures the lowest contrast (contrast sensitivity) to see red, green, blue and grey letters.
Change in Color Naming Accuracy on Cone Contrast Color Naming test (CCNT) | This test will occur prior to the intervention (Meibomian gland expression) and immediately after this intervention.
  This computer test measures the accuracy of naming (number correct) low contrast red, green, blue and grey letters.

OTHER OUTCOMES:
Change in High Contrast Visual Acuity | This test will occur prior to the intervention (Meibomian gland expression) and immediately after this intervention.
  The Precision Vision, Inc. Super Vision Chart will be used to measure visual acuity (smallest black letters on a white background that can be seen).
Change in Small Letter Contrast Sensitivity | This test will occur prior to the intervention (Meibomian gland expression) and immediately after this intervention.
  The Precision Vision, Inc. Super Vision Chart will be used to measure the lowest contrast (contrast sensitivity) which can be seen using small (20/25) letters.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Rabin, OD, PhD, Study Chair — University of the Incarnate Word
Locations (1):
- University of the Incarnate Word Rosenberg School of Optometry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Share IPD will facilitate data analysis and understanding for current and future research. We will share outcome and results and potentially present to local, national, and international faculty during conferences.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available upon conclusion of the study and for approximately 1 year.

REFERENCES:
- [Background] Gao Y, Liu R, Liu Y, Ma B, Yang T, Hu C, Qi H. Optical quality in patients with dry eye before and after treatment. Clin Exp Optom. 2021 Jan;104(1):101-106. doi: 10.1111/cxo.13111. PMID 32618024
- [Background] Szczotka-Flynn LB, Maguire MG, Ying GS, Lin MC, Bunya VY, Dana R, Asbell PA; Dry Eye Assessment and Management (DREAM) Study Research Group. Impact of Dry Eye on Visual Acuity and Contrast Sensitivity: Dry Eye Assessment and Management Study. Optom Vis Sci. 2019 Jun;96(6):387-396. doi: 10.1097/OPX.0000000000001387. PMID 31116166
- [Background] Narayanan S, Miller WL, Prager TC, Jackson JA, Leach NE, McDermott AM, Christensen MT, Bergmanson JP. The diagnosis and characteristics of moderate dry eye in non-contact lens wearers. Eye Contact Lens. 2005 May;31(3):96-104. doi: 10.1097/01.icl.0000140907.45705.e2. PMID 15894874
- [Background] Thulasi P, Djalilian AR. Update in Current Diagnostics and Therapeutics of Dry Eye Disease. Ophthalmology. 2017 Nov;124(11S):S27-S33. doi: 10.1016/j.ophtha.2017.07.022. PMID 29055359
- [Background] Yeh TN, Lin MC. Meibomian Gland Contrast Sensitivity and Specificity in the Diagnosis of Lipid-deficient Dry Eye: A Pilot Study. Optom Vis Sci. 2021 Feb 1;98(2):121-126. doi: 10.1097/OPX.0000000000001636. PMID 33534375